CLINICAL TRIAL: NCT06337240
Title: Pelvic Floor Exercises Versus Pilates on Urinary Incontinance in Chronic Obstructive Pulmonary Disease
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Ayman, physiotherapist, Cairo University
Other Study IDs: pelvic floor exercise
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic floor exercises on COPD patients: 30 COPD female patients with urinary incontinence will receive pelvic floor exercises.
  Interventions: Other: Pelvic floor on COPD patients; Other: Pilates exercises on COPD patients

INTERVENTIONS:
Other: Pelvic floor on COPD patients — Group A (study group) :
  This group will include 30 COPD patients with urinary incontinence , who will receive pelvic floor exercise for 3 days a week for a total of 3 months.
Other: Pilates exercises on COPD patients — Group B (study group):
  This group will include 30 COPD patients with urinary incontinence , who will receive pilates for 3 days a week for a total 3 months.

SUMMARY:
The aim of the study is To compare between the effect of both pelvic floor and Pilates exercises on urinary incontinences in COPD patients.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is defined as loss of bladder control and is characterized by the complaint of any involuntary leakage of urine UI is an important individual and social problem, in that it is associated with worse health-related quality of life (HRQoL) in subjects with chronic obstructive pulmonary disease. Although UI is not a life-threatening condition, it is common and can have numerous negative psychological, social, and economical effects. Women with UI in the general population have higher levels of depression, anxiety and stress, poor sleep quality and significantly lower HRQL Additionally, long term UI may result in absence from work, increased healthcare costs, social isolation and physical inactivity which is common from the early stages of the COPD due to dyspnea. Furthermore, inactivity is associated with risk of hospital admissions and is a strong predictor for mortality. The combination of UI and COPD may therefore result in a double risk factor in terms of exercise avoidance and the subsequent negative consequences of inactivity.

As it could be concluded that urinary incontinence is a trouble problem that can change the life of COPD patients and therapy attempts to prevent it or control it will be appreciated, taking in consideration that all people nowadays prefer to choose the most safe method of their conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD & Urinary incontinence
* Stable with moderate to severe COPD
* Their ages will range from fifty years old.
* All patients will be clinically stable.

Exclusion Criteria:

* Gynecologic surgery ( 6 months prior to study)
* Current urinary tract infection
* Uncontrolled Diabetes Mellitus
* Diagnosed with psychiatric or depressive disorder
* Existing arterial aneurysm.
* Clinical signs of unstable cardiac event (eg, congestive heart failure),
* Severe arterial hypertension,
* Neurological disorders that will affect pelvic floor muscles.
* Acute COPD exacerbation within the last 4 weeks.
* Any need for supplemental oxygen.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 60 females in the study
Study Population: Group A (study group) :
  This group will include 30 COPD patients with urinary incontinence , who will receive pelvic floor exercise for 3 days a week for a total of 3 months.
  Group B (study group):
  This group will include 30 COPD patients with urinary incontinence , who will receive Pilates for 3 days a week for a total 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2024-07-02 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence (1 Hour and 24- Hour pad test) | 3 months
  Pad testing is a non-invasive method of detecting and quantifying severity of urine leakage in men or women.
Incontinence severity index: | 3 months
  Incontinence Severity Index (ISI), consisting of two questions regarding frequency (four levels) and amount (three levels) of leakage. The validity of the ISI has been demonstrated for different types of UI and has received the highest recommendation from the 2nd and 3rd International Consultation on Incontinence

SECONDARY OUTCOMES:
Urinary incontinence quality of life questionnaire (I-QOL) | 3 months
  Incontinence Quality of Life (I-QOL), a condition-specific instrument designed to measure the QOL effects of UI in women. The I-QOL contains 22 items with a 5-point Likert-type response scale yielding a total score and three subscale scores (i.e., avoidance and limiting behaviors, psychosocial impacts, and social embarrassment) with good to excellent test-retest reliability
Cough symptoms score | 3 months
  its reliability and treatment response have been confirmed The CSS is a two-part questionnaire referring to daytime and night-time symptoms. Based on the frequency, intensity and influence of cough on daily activities and sleep, cough symptoms are scored from 0 to 5, with 0 indicating no cough and 5 indicating the most severe cough
Cough symptoms questionnaire | 3 months
  It is a questionnaire consisting of 19 items, including 8 physical items, 7 psychological items and 4 social items. Each item is rated according to the frequency of occurrence with a score ranging from 1 to 7. The regional score is the sum of items scored divided by the items (score 1-7) in each area; the total score is the sum of the regional scores.The lower the score, the more serious the impact of chronic cough un quality of life
The COPD Assessment Tool (CAT) | 3 months
  This COPD-specific questionnaire evaluates the overall burden in subjects with COPD using 8 different questions. Each question can be scored from 0 points (not impaired) to 5 points (maximally impaired). Accordingly, the total score can range from 0 to 40 points, with higher scores reflecting greater burden of the disease.
  CAT questionnaire consisting of eight questions regarding cough, phlegm, chest tightness, breathlessness during activities, activity limitations at home, confidence in leaving home, sleep and energy. The scoring range of each item is between 0 and 5, with a maximum score of 40.
  According to the total CAT scores, the patients were included in the following stages:
  Stage 1: <10 Stage 2: 10-20 Stage 3: >20 Stage 4: >30(

CONTACTS AND LOCATIONS:
Overall Officials: Donia El Masry, Doctorate, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020